CLINICAL TRIAL: NCT00044889
Title: A Phase II, Open-Label Study of Clofarabine in Adult Patients With Refractory or Relapsed Acute Myelogenous Leukemia
Brief Title: Phase II Study of Clofarabine in Adult Patients With Refractory or Relapsed Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLO221
Record Dates: First submitted 2002-09-06; First posted 2002-09-09 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Acute Myelogenous Leukemia
Keywords: CLO221; clolar
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Clofarabine; Dosage Forms

INTERVENTIONS:
Drug: clofarabine (IV formulation)

SUMMARY:
Clofarabine (injection) is approved by the Food and Drug Administration (FDA) for the treatment of pediatric patients 1 to 21 years old with relapsed acute lymphoblastic leukemia (ALL) who have had at least 2 prior treatment regimens.

This is a single arm, open-label, Phase II study of CLOFARABINE in adult patients with refractory or relapsed acute myelogenous leukemia (AML). Qualified patients must be refractory to one or two induction regimens, or have relapsed < one year from the date of confirmation of the initial complete remission (CR). There will be two phases in this study - an Induction phase and a Consolidation phase.

ELIGIBILITY:
Inclusion Criteria:

* note: For inclusion and exclusion criteria, a regimen is defined as including Induction, Consolidation, and Maintenance therapies.
* Diagnosis of AML according to FAB classification
* Must not be eligible for therapy of higher curative potential, and must be in first or subsequent relapse and/or refractory
* A Karnofsky Performance Status (KPS) of greater than or equal to 60.
* If female of childbearing potential, patients must have a negative serum or urine pregnancy test within 7 days of study enrollment. Men and women with reproductive potential must use as an effective contraceptive method while enrolled in the study. Patients must have contraceptive and/or fertility counseling prior to entering the study, i.e., information on sperm banking, etc.
* Signed, written informed consent.
* Ability to comply with study procedures and follow-up examinations.
* Adequate organ function as indicated by specific laboratory values (defined in the protocol), obtained within two weeks prior to registration.
* Classified as AML FAB M3 (Acute Promyelocytic leukemia) and have been treated with at least 2 regimens (a retinoic acid containing regimen and an arsenic trioxide containing regimen) before being considered for this study.

Exclusion Criteria:

* note: For inclusion and exclusion criteria, a regimen is defined as including Induction, Consolidation, and Maintenance therapies.
* Received previous treatment with CLOFARABINE.
* Received more than two previous induction regimens or cycles for the treatment of AML.
* Relapsed > 1 year.
* Have an active, uncontrolled systemic infection considered opportunistic, life threatening, or clinically significant at the time of treatment.
* Are pregnant or lactating.
* Have psychiatric disorders that would interfere with consent, study participation or follow-up.
* Are receiving any other chemotherapy or corticosteroids. Patients must be off previous therapy for at least two weeks and must have recovered from acute toxicity of all previous therapy prior to enrollment.
* Have any other severe concurrent disease.
* Have symptomatic CNS involvement.
* Have chronic myelogenous leukemia (CML) in lymphoid blast crisis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-05; Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (12):
- United States (12):
  - Los Angeles, California
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Chicago, Illinois
  - St Louis, Missouri
  - Omaha, Nebraska
  - Buffalo, New York
  - Durham, North Carolina
  - Memphis, Tennessee
  - Houston, Texas
  - Norfolk, Virginia
  - Seattle, Washington